CLINICAL TRIAL: NCT00409643
Title: A Randomized, Double-blind, Multicenter, Multifactorial, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Valsartan (160 mg and 320 mg) and Amlodipine (10 mg) Combined and Alone in Hypertensive Patients
Brief Title: Safety and Efficacy of Valsartan and Amlodipine Combined and Alone in Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAA489A2307
Record Dates: First submitted 2006-12-07; First posted 2006-12-11 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: HYPERTENSION, VALSARTAN, AMLODIPINE, high blood pressure
MeSH Terms: conditions — Hypertension | interventions — Amlodipine, Valsartan Drug Combination; Valsartan; Amlodipine

INTERVENTIONS:
Drug: valsartan+amlodipine combination
Drug: valsartan
Drug: amlodipine

SUMMARY:
This trial will compare valsartan and amlodipine combination therapies to valsartan and amlodipine monotherapy,and placebo for treating patients with hypertension

ELIGIBILITY:
Inclusion Criteria:

* Outpatients 18 years and older.
* Male or female patients are eligible. Female patients must be either post-menopausal for one year or surgically sterile, or using effective contraceptive methods such as barrier method with spermicide or an intra-uterine device. Hormonal contraceptive use is disallowed.
* Patients with essential diastolic hypertension measured by calibrated standard aneroid or mercury (preferable) sphygmomanometer. Patients must have a MSDBP > 90 mmHg and < 110 mmHg at Visit 1 (week -4 to -2), and a MSDBP > 95 mmHg and < 110 mmHg at Visit 2 (week 0).
* Patients must have an absolute difference of > 10 mmHg in their average sitting diastolic blood pressure between Visits 1 and 2.
* Patients who are eligible and able to participate in the study, and who consent to do so after the purpose and nature of the investigation has been clearly explained to them (written informed consent).

Exclusion Criteria:

* Severe hypertension (MSDBP 110 mmHg and/or MSSBP 180 mmHg) at anytime.
* Inability to discontinue all prior antihypertensive medications safely for a period of 14 weeks.
* Known Keith-Wagener grade III or IV hypertensive retinopathy.
* History of hypertensive encephalopathy or cerebrovascular accident at anytime prior to Visit 0 (week -6 to -4).
* Transient ischemic cerebral attack during the last 12 months prior to Visit 0 (week -6 to -4).
* Evidence of a secondary form of hypertension, such as coarctation of the aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing Disease, pheochromocytoma, polycystic kidney disease etc.
* Type 1 diabetes mellitus.
* Type 2 diabetes mellitus with poor glucose control as defined by fasting glycosylated hemoglobin (HbA1c) >8% at Visit 1 (week -4 to -2).
* Administration of any agent indicated for the treatment of hypertension within a minimum 4 weeks prior to randomization into the study (Visit 2, week 0), with the permitted exception of those anti-hypertensive medications requiring tapering down commencing at Visit 0 (week -6 to -4).
* Known or suspected contraindications, including history of allergy to angiotensin receptor blockers or calcium channel blockers.
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1259 (Actual)
Dates: Start 2004-01; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline (Visit 2) in mean sitting diastolic blood pressure at trough (endpoint-Week 8).

SECONDARY OUTCOMES:
Change from baseline (Visit 2) in mean sitting systolic blood pressure at trough (endpoint-Wk 8)
Change from baseline (Visit 2) in standing diastolic and systolic blood pressure at trough(endpoint-Wk 8)
Sitting and standing pulse

CONTACTS AND LOCATIONS:
Overall Officials: Novartis pharmaceuticals, Study Chair — Sponsor GmbH
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Sites in Germany, Germany, Germany